CLINICAL TRIAL: NCT03275350
Title: Comparing Treatments for HIV-Infected Opioid Users in an Integrated Care Effectiveness Study (CHOICES) Scale-Up
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Johns Hopkins University (Other); University of Kentucky (Other); Jackson Health System (Other); Tarzana Treatment Centers (Other); Ruth M. Rothstein CORE Center (Other)
Responsible Party: Principal Investigator, P. Todd Korthuis, MD, Professor of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clinical Trials Network-0067
Record Dates: First submitted 2017-08-28; First posted 2017-09-07 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Opioid-use Disorder; Hiv
MeSH Terms: conditions — Opioid-Related Disorders; Acquired Immunodeficiency Syndrome | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- XR-NTX (Active Comparator): Extended-release naltrexone
  Interventions: Drug: Naltrexone Injectable Suspension
- TAU (Active Comparator): Treatment as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Drug: Naltrexone Injectable Suspension — Six monthly injections of extended-release naltrexone
  Arms: XR-NTX
Other: Treatment as usual — Standard treatment for opioid use disorder provided at each HIV clinic
  Arms: TAU

SUMMARY:
The Primary Objective of this study is to compare the effectiveness of HIV clinic-based extended-release Naltrexone (XR-NTX) in decreasing substance use and increasing HIV viral suppression in HIV-infected participants with opioid use disorder to Treatment as Usual in this population.

DETAILED DESCRIPTION:
The CTN-0055 CHOICES pilot study demonstrated the feasibility of extended-release naltrexone (XR-NTX) for treatment of opioid use disorder in HIV primary care. The CTN-0067 CHOICES scale-up study builds on lessons learned from the pilot and uses the Consolidated Framework for Implementation Research to advance understanding of XR-NTX adoption in HIV primary care clinics. The study is an open-label, randomized, comparative effectiveness trial of office-based XR-NTX for 24 weeks (6 monthly injections) versus treatment as usual (TAU) in HIV-infected participants with untreated opioid use disorder. Each participant will be engaged in the overall study for 25 to 28 weeks, depending on the speed of screening and enrollment procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years old
* Participant has provided written informed consent and HIPAA for medical record abstraction
* Participant meets Diagnostic and Statistical (DSM)-5 criteria for moderate or severe opioid use disorder
* Willing to be randomized to antagonist-based therapy or TAU for treatment of opioid use disorder
* Has an HIV viral RNA count of greater than 200 copies/ml (not clinically suppressed)
* Willing to establish ongoing HIV care at the site if not already receiving ongoing care
* If female, willing to take at least one evidence-based measure to avoid becoming pregnant

Exclusion Criteria:

* Participant has a serious medical, psychiatric, or substance use disorder that, in the opinion of the study physician, would make participation hazardous to the participant, compromise study findings, or prevent participant from completing the study. Examples include:
* Acutely life-threatening medical illnesses (e.g., active opportunistic infection, uncompensated heart failure, end-stage liver disease, acute hepatitis and moderate to severe renal impairment) as assessed by medical history, review of symptoms, physical exam and/or laboratory assessments
* Severe, inadequately treated mental health disorder (e.g., active psychosis, uncontrolled manic-depressive illness) as assessed by history and/or clinical interview
* Suicidal or homicidal ideation requiring immediate attention
* Participant has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) liver enzymes greater than five times the upper limit of normal on screening phlebotomy
* Participant has an international normalized ratio (INR) > 1.5 or platelet count <100k
* Participant has a known allergy or sensitivity to naloxone, naltrexone, polyactide-co-glycolide, carboxymethylcellulose, or other components of the Vivitrol diluent
* Anticipate undergoing surgery during study participation
* Have chronic pain requiring ongoing pain management with opioid analgesics
* If female, currently (at time of consent) pregnant or breastfeeding or planning on conceiving in the coming months
* Body habitus that, in the judgment of the study physician, precludes safe intramuscular injection on XR-NTX (e.g., excess fat tissue over the buttocks)
* Received methadone of buprenorphine maintenance therapy for treatment of opioid dependence in the 4 weeks prior to screening
* Have taken an investigational drug in another study within 30 days of study consent
* Have had treatment with XR-NTX for opioid or alcohol dependence in the 4 weeks prior to consent
* Are currently in jail, prison or have a pending legal action which may prevent an individual from completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Tarzana Treatment Centers, Tarzana, California
  - Jackson Memorial Hospital, Miami, Florida
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - University of Kentucky Bluegrass Care Clinic, Lexington, Kentucky
  - Johns Hopkins University, Bartlett Specialty Clinic, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Foot C, Korthuis PT, Tsui JI, Luo SX, Chan B, Cook RR. Associations between stimulant use and return to illicit opioid use following initiation onto medication for opioid use disorder. Addiction. 2024 Jan;119(1):149-157. doi: 10.1111/add.16334. Epub 2023 Sep 15. PMID 37712113
- [Derived] Hoffman KA, Baker R, Fanucchi LC, Lum PJ, Kunkel LE, Ponce Terashima J, McCarty D, Jacobs P, Korthuis PT. Perspectives on extended-release naltrexone induction among patients living with HIV and opioid use disorder: a qualitative analysis. Addict Sci Clin Pract. 2021 Nov 10;16(1):67. doi: 10.1186/s13722-021-00277-z. PMID 34758887

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended-release Naltrexone (XR-NTX): Extended-release naltrexone
  Naltrexone Injectable Suspension: Six monthly injections of extended-release naltrexone
- Treatment as Usual (TAU): Treatment as usual
  Treatment as usual: Standard treatment for opioid use disorder provided at each HIV clinic
Period: Overall Study
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Started | 55 | 59
Completed | 47 | 51
Not Completed | 8 | 8
Not completed — Lost to Follow-up | 4 | 6
Not completed — Death | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Incarcerated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 55 | 59 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (10.8) | 46 (11.5) | 47 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 32 | 39 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 46 | 54 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 34 | 64
  White | 19 | 23 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8
HIV Viral Load [Mean (Standard Deviation); unit: log10 copies/mL] | 4.0 (0.9) | 4.0 (1.1) | 4.0 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HIV Viral Suppression, Missing Imputed as Unsuppressed
Description: HIV-1 RNA <200 copies/ml
Time Frame: 12 weeks and 24 weeks
Population: Non-inferiority analyses of HIV viral suppression by treatment arm Intent to Treat Group Missing imputed as unsuppressed
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 55 | 59
Participants
  12 Weeks | 23 | 21
  24 Weeks | 29 | 29

2. Primary Outcome: Number of Participants With HIV Viral Suppression, Complete Case
Description: HIV-1 RNA <200 copies/ml
Time Frame: 12 weeks and 24 weeks
Population: Non-inferiority analyses of HIV viral suppression by treatment arm Complete case: Includes 81 participants with non-missing viral load data at 12 and 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 42
Participants
  12 Weeks | 23 | 19
  24 Weeks | 26 | 26

3. Primary Outcome: Number of Participants With HIV Viral Suppression, Per-protocol
Description: HIV-1 RNA <200 copies/ml
Time Frame: 12 weeks and 24 weeks
Population: Non-inferiority analyses of HIV viral suppression by treatment arm Missing as unsuppressed Per-protocol population includes 69 participants who received at least one dose of their assigned study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 26 | 43
Participants
  12 weeks | 11 | 16
  24 weeks | 15 | 23

4. Secondary Outcome: Veterans Aging Cohort Study (VACS) Index
Description: Absolute value of participant VACS Index at baseline and 24 weeks
  Veterans Aging Cohort Study Index Minimum value: 0 Maximum value: 164 A higher score means a worse outcome.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 55 | 59
score on a scale
  Baseline | 65.1 (18.1) | 68.4 (24.7)
  24 Weeks | 54.4 (20.7) | 63.5 (25.4)

5. Secondary Outcome: CD4 Count
Description: Cluster of Differentiation 4
  Absolute value of CD4 count at baseline and 24 weeks.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: cells/mm3
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 55 | 59
cells/mm3
  Baseline | 380.7 (248.2) | 439.8 (336.6)
  24 Weeks | 459.1 (249.1) | 505.1 (349.1)

6. Secondary Outcome: Engagement in HIV Care: Antiretroviral Therapy Prescribed
Description: Absolute value of participants prescribed ART at baseline and within 24 weeks following randomization. Each individual can be scored 0 (not prescribed ART) or 1 (prescribed ART) at both baseline and follow-up, after which his or her outcome score will be the follow-up score minus the baseline score. Outcomes will be analyzed via rank-based methods such as Wilcoxon rank-sum tests.
Time Frame: Baseline and 24 weeks
Population: Number analyzed at 24 weeks lower than baseline due to study retention and availability of data.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 55 | 59
Participants
  Baseline | 37 | 46
  24 Weeks: number analyzed (Participants) | 48 | 52
  24 Weeks | 45 | 43

7. Secondary Outcome: Engagement in HIV Care: 100% Antiretroviral Therapy Adherence
Description: Number of participants taking 100% of prescribed ART doses in the past month at 24 weeks for those prescribed ART at any point during the 24 week trial (proportion; self-reported medication adherence measure). Chi-squared test comparing proportion to treatment assignment, for those prescribed ART.
Time Frame: 24 weeks
Population: This outcome measure is based on participant self-report. As such, fewer participants provided data for this outcome measure than other measures where data was obtained through pharmacy or clinic attendance logs.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 45 | 45
Participants | 16 | 13

8. Secondary Outcome: Number of Participants With at Least 1 HIV Care Visit in Past 12 Weeks
Description: At least 1 HIV care visit in past 12 weeks
Time Frame: 24 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 52 | 58
Participants | 31 | 29

9. Secondary Outcome: Number of Participants Who Had Unprotected Sex in Past 30 Days
Description: Past 30 day unprotected sex, as measured by the Risk Assessment Battery at baseline and week 24 (binary; self-report).
Time Frame: Baseline and 24 weeks
Population: Those reporting no sex are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 27 | 30
Participants
  Baseline | 15 | 16
  24 Weeks: number analyzed (Participants) | 15 | 21
  24 Weeks | 9 | 9

10. Secondary Outcome: Number of Participants With Multiple Sex Partners in Past 30 Days
Description: Past 30 day multiple sex partners, as measured by the Risk Assessment Battery at baseline and week 24 (binary; self-report).
Time Frame: Baseline and 24 weeks
Population: Two or more sex partners during past month, those reporting no sex partners are excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 25 | 26
Participants
  Baseline | 10 | 6
  24 Weeks: number analyzed (Participants) | 12 | 21
  24 Weeks | 5 | 6

11. Secondary Outcome: Engagement in HIV Care: Quality of Life
Description: Past 30 day health-related quality of life as measured by the EQ-5D questionnaire at baseline and week 24.
  Minimum value: 0 Maximum value: 100 Higher scores mean a better outcome
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 55 | 59
score on a scale
  Baseline | 58 (19.1) | 64.3 (17.6)
  24 Weeks | 67.9 (21.2) | 71.2 (19.1)

12. Secondary Outcome: Average Number of Self-Reported Days of Opioid Use in Last 30 Days
Description: Average number of days of opioid use between baseline and 24 weeks, measured by the Timeline Follow-Back (count; self-report), will be used to compare opioid use by treatment group. Confirmatory analysis will assess opioid use by the average number of days of opioid use in the last 30 days of the study (by Addiction Severity Index-lite; count; self-report) and the number of monthly urine drug screen (UDS) negative for opioids between baseline and 24 weeks (count; laboratory data).
Time Frame: Between baseline and 24 weeks
Population: Per-protocol population includes participants who received at least one dose of their assigned study medication.
Measure: Mean (Full Range); unit: days
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 55 | 59
days
  Intent-to-treat | 11.73 [0 to 30] | 14.81 [0 to 30]
  Per-protocol: number analyzed (Participants) | 26 | 43
  Per-protocol | 6.02 [0 to 30] | 13.58 [0 to 30]

13. Secondary Outcome: Number of Participants Who Test Positive for Opioids at 24 Weeks
Description: Number and percent of participants with UDS positive for opioids at 24 weeks.
Time Frame: 24 weeks
Population: Per-protocol population includes participants who received at least one dose of their assigned study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
Number analyzed (Participants) | 55 | 59
Participants
  Intent-to-treat | 34 | 40
  Per-protocol: number analyzed (Participants) | 26 | 43
  Per-protocol | 10 | 30

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Extended-release Naltrexone (XR-NTX) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 2/55 | 1/59
Serious Adverse Events (participants affected / at risk) | 5/55 | 7/59
Other Adverse Events (participants affected / at risk) | 11/55 | 7/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended-release Naltrexone (XR-NTX) (N=55) | Treatment as Usual (TAU) (N=59)
Infections (Infections and infestations) | 2 (2) | 3 (3)
Psychiatric disorders (Psychiatric disorders) | 2 (2) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vascular disorders (Vascular disorders) | 1 (1) | 0 (0)
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended-release Naltrexone (XR-NTX) (N=55) | Treatment as Usual (TAU) (N=59)
Infections (Infections and infestations) | 2 (2) | 5 (5)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) | 0 (0)
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 2 (2) | 1 (1)
Nervous system disorders (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT03275350/Prot_SAP_000.pdf